CLINICAL TRIAL: NCT06383780
Title: A Randomized, Controlled, Multicenter Clinical Study Comparing the Efficacy of Pembrolizumab in Combination With Nab-TPC Regimen Versus the GP Regimen in the First-Line Treatment of Nasopharyngeal Carcinoma With Bone Metastases.
Brief Title: Tislelizumab in Combination With GP or TPC Regimen for the Treatment of Nasopharyngeal Carcinoma With Bone Metastasis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: XIANG YANQUN (Other)
Responsible Party: Sponsor-Investigator, XIANG YANQUN, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-901-01
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma With Bone Metastasis; immunochemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: Active Comparator:Drug:GP（Gemcitabine combined with cisplatin）regimen combined with Tislelizumab Experimental:Drug：TPC（cisplatin, nab-paclitaxel and capecitabine）regimen combined with Tislelizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP combined with Tislelizumab (Active Comparator): Gemcitabine combined with cisplatin regimen combined with Tislelizumab
  Interventions: Drug: GP combined with Tislelizumab
- TPC combined with Tislelizumab (Experimental): cisplatin, nab-paclitaxel and capecitabine regimen combined with Tislelizumab
  Interventions: Drug: TPC combined with Tislelizumab

INTERVENTIONS:
Drug: GP combined with Tislelizumab — Gemcitabine combined with cisplatin regimen combined with Tislelizumab
  Arms: GP combined with Tislelizumab
Drug: TPC combined with Tislelizumab — cisplatin, nab-paclitaxel and capecitabine regimen combined with Tislelizumab
  Arms: TPC combined with Tislelizumab

SUMMARY:
This is a prospective, open-label phase III clinical trial evaluating the efficacy and safety of the GP（Gemcitabine combined with cisplatin） regimen in combination with Tislelizumab versus the TPC（cisplatin, nab-paclitaxel and capecitabine）regimen in combination with Tislelizumab for the first-line treatment of Nasopharyngeal Carcinoma patients With Bone Metastasis.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of the GP regimen combined with Tislelizumab compared to the TPC regimen combined with Tislelizumab in the treatment of advanced first-line bone metastatic nasopharyngeal carcinoma patients in high-risk nasopharyngeal carcinoma areas through a prospective, open-label phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years.
2. Histology or cytology confirmed nasopharyngeal carcinoma.
3. Metastatic nasopharyngeal carcinoma of bone that is not suitable for local or radical therapy.
4. Distant bone metastases confirmed by imaging (two images) or pathology (plus one image) (AJCC 8th, stage IVB), except for isolated local invasion of the base bone of the skull.
5. With or without metastases from other organs, but lesions may be non-measurable distant organ metastases or lymph node lesions (as assessed by RECIST 1.1).
6. Bone metastases may contain soft tissue components of osteolytic lesions.
7. Patients have not previously received systemic therapy for advanced or metastatic disease, and prior induction chemotherapy, concurrent chemoradiotherapy, or adjuvant chemotherapy must have been completed more than 6 months prior to enrollment. Previous radiotherapy or concurrent chemoradiotherapy should also be completed more than 6 months prior to enrollment.
8. Expected survival ≥ 3 months.
9. According to the Eastern Cooperative Oncology Group (ECOG) criteria, the performance status score is 0 or 1.
10. Good organ function:Hemoglobin > 8.0 g/dl; Absolute neutrophil count (ANC) >1,500/mm3; Platelet count> 100,000/μl; Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase and glutamate aminotransferase < 2.5 ULN (upper limit of normal), (alanine aminotransferase and aspartate aminotransferase < 5 ULN in patients with liver metastases), alkaline phosphatase< 4 ULN;Prothrombin time (PT) international normalized ratio/prothrombin time (PTT) < 1.5 ULN, serum muscle；Anhydride< 1.5ULN.
11. Willing and able to comply with planned visits, treatment plans, laboratory tests, and other research procedures.

Exclusion Criteria:

1. Patients with osteo-oligometastatic nasopharyngeal carcinoma.
2. Previous history of severe hypersensitivity to any component of other monoclonal antibodies or tislelizumab monoclonal mab.
3. Patients have ≥ 1 metastatic organs or lymph node lesions that can be measured (assessed according to RECIST 1.1)
4. No definitive surgical and/or radiotherapy for spinal cord compression, or for previously diagnosed and treated spinal cord compression, no evidence that the disease was clinically stable for ≥ 2 weeks prior to enrollment.
5. Poorly controlled pleural effusion, pericardial effusion, or ascites requiring frequent drainage. Patients with indwelling catheters, such as PleurX ® catheters, are allowed to participate.
6. Poorly controlled tumor-related pain. Patients requiring analgesic therapy must receive a stable dose before enrolling in the study. Patients who are candidates for palliative radiation therapy (e.g., bone metastases or metastases leading to nerve damage) should be treated prior to enrollment Lesions are treated. Prior to enrollment, if appropriate, consideration should be given to the need for further growth that may result in functional deficits or intractable pain (e.g., For example, asymptomatic metastases currently not associated with spinal cord compression) are treated locally-regionally.
7. Poorly controlled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium> 12 mg/dL or corrected serum calcium higher than ULN)
8. Malignancy with malignancies other than nasopharyngeal carcinoma within 5 years prior to enrollment, with negligible risk of metastasis or death (e.g., expected 5-year OS>90%) and expected radical results after treatment (e.g., adequately treated cervix).

   Localized cancer, basal or squamous cell skin cancer, localized prostate cancer treated for radical purposes, surgical treatment for radical purposes Ductal carcinoma in situ).
9. History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis related to antiphospholipid syndrome, Wegener's granuloma disease, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with autoimmune-related hypothyroidism receiving stable dose thyroid hormone replacement therapy were eligible to participate in this study. Patients with type 1 diabetes who are controlled after receiving a stable insulin regimen are eligible to participate in this study.
10. Receiving systemic immunostimulating drugs (including but not limited to interferon or IL-2) within 4 weeks prior to enrollment or within 5 half-lives of the drug (whichever is shorter).
11. Receiving systemic corticosteroids (> 10 mg/d prednisone equivalent) or other systemic immunosuppressants (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide and antibody) within 2 weeks prior to enrollment Tumor necrosis factor drugs [anti-TNF]). Topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are permitted. Patients receiving acute low-dose systemic immunosuppressive agents (e.g., a single dose of dexamethasone for nausea) can be considered after a comprehensive discussion to decide whether to enroll in the study. Prophylactic steroids may be used in patients requiring baseline and follow-up MRI tumor evaluation who have had a previous allergic reaction to intravenous contrast.
12. Patients who have previously undergone allogeneic bone marrow transplantation or have previously undergone solid organ transplantation.
13. History of idiopathic pulmonary fibrosis, drug-induced pneumonia, organic pneumonia (ie, bronchiolitis obliterans), history of idiopathic pneumonia or chest CT scan showing evidence of active pneumonia at screening.
14. Active infection, including tuberculosis (clinical diagnosis includes clinical history, physical examination and imaging findings, and TB examination according to local medical practice), hepatitis B (known HBV surface antigen (HBsAg)), hepatitis C, or human immunodeficiency virus (HIV antibody positive). Patients with previous or cured HBV infection (defined as hepatitis B core antibody [anti-HBc] positive and HbsAg-negative) are eligible to participate in this study only if they are HBV DNA negative (HBV DNA ˂1000cps/ml). Patients with positive hepatitis C (HCV) antibodies have only polymerase chain reaction (PCR) that is HCV RNA negative is eligible to participate in this study.
15. Clinically significant underlying medical conditions (e.g., dyspnea, pneumonia, pancreatitis, poorly controlled diabetes, active or poorly controlled infections, drugs, or alcohol) that the investigator believes may affect study drug administration and protocol adherence abuse, or mental illness).
16. Presence of severe neurological or psychiatric disorders, including dementia and seizures.
17. Accompanied by NCI-CTCAE ≥ grade 2 peripheral neuropathy.
18. Pregnant or lactating female patients.
19. Major cardiovascular diseases, such as New York Heart Association heart disease (grade II or higher, see Appendix 6), myocardial infarction within 3 months prior to enrollment, unstable arrhythmias or unstable angina. Known to have coronary artery disease, not satisfied Patients with standard congestive heart failure or left ventricular ejection fraction < 50% must be treated with an optimized stable medical regimen as determined by the treating physician, and if appropriate, a cardiologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival rate | up to 3 years

SECONDARY OUTCOMES:
Overall survival | up to 3 years
incidence of adverse events | up to 3 years
  safety
rate of skeletal-related events | up to 3 years
Biomarker response (EBV-DNA, bone metabolic markers) | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The diagnosis, treatment regimen, toxicity and followup data will be shared once every year through email, phone or meeting.